CLINICAL TRIAL: NCT05451472
Title: Evalution of Thyroid Functions in Hemodialysis Children in Sohag University Hospital
Brief Title: Evluation of Thyroid Functions in Hemodialysis Childern in Sohag University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Michael Rafat Helmi, resident doctor at pediatric department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: soh-22-06-09
Record Dates: First submitted 2022-06-20; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Chronic Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Thyroid Function Tests; Blood Cell Count; Blood Urea Nitrogen; Liver Function Tests; Blood Gas Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pediatric group (Experimental)
  Interventions: Diagnostic Test: thyroid function tests; Diagnostic Test: complete blood count; Diagnostic Test: serum creatinine; Diagnostic Test: blood urea; Diagnostic Test: serum electrolyte; Diagnostic Test: serum calcium; Diagnostic Test: serum phosphorus; Diagnostic Test: parathyroid hormone level; Diagnostic Test: liver function test; Diagnostic Test: arterial blood gases; Diagnostic Test: complete urine analysis

INTERVENTIONS:
Diagnostic Test: thyroid function tests — Thyroid function tests:thyroid stimulating hormone (TSH), total thyroxine (T4), free thyroxine (FT4), total triiodothyronine (T3), and free triiodothyronine (FT3)
Diagnostic Test: complete blood count — complete blood count
Diagnostic Test: serum creatinine — serum creatinine
Diagnostic Test: blood urea — blood urea
Diagnostic Test: serum electrolyte — serum electrolyte
Diagnostic Test: serum calcium — serum calcium
Diagnostic Test: serum phosphorus — serum phosphorus
Diagnostic Test: parathyroid hormone level — parathyroid hormone level
Diagnostic Test: liver function test — ALT_AST_Total biliruin_total protein _serum albumin
Diagnostic Test: arterial blood gases — PH_PCO2_PO2_HCO3_base deficit
Diagnostic Test: complete urine analysis — complete urine analysis

SUMMARY:
Thyroid gland and its hormones play an important role in organ development and the homeostatic control of many physiological mechanisms such as body growth and energy expenditure. The two main thyroid hormones are triiodothyronine (T3) and thyroxine (T4) affect renal development and metabolism so any impairment in thyroid functions lead to or aggravate kidney diseases.

On the other hand, kidneys play an important role in the thyroid metabolism as it normally contributes to the clearance of iodide, primarily by glomerular filtration. Among patients with renal failure, there is diminished iodide excretion and an increase in plasma inorganic iodide, which results in increased uptake of the iodide by the thyroid gland. Increases in total body inorganic iodide can potentially block thyroid hormone production (the Wolff-Chaik off effect). Such a change may explain the slightly higher frequency of goiter and hypothyroidism in patients with chronic kidney diseases.

The kidneys affect the hypothalamic pituitary-thyroid axis, so any impairment in kidney functions leads to disturbed thyroid physiology. All levels of the hypothalamic-pituitary-thyroid axis may be involved, including alterations in hormone production, distribution, and excretion.

End stage renal disease (ESRD) and hemodialysis (HD) affect the levels of all thyroid hormones. The earliest and the most common thyroid function abnormality in patients with ESRD on HD is low T3 level (especially total T3 than free T3). This is called 'low T3 syndrome. The prevalence of subclinical hypothyroidism has been reported to be much higher in patients with ESRD on HD than in the general population.

Due to similarity of signs and symptoms, sometimes it is difficult to identify subjects with ESRD also has hypothyroidism; therefore, different studies have been carried out to establish the incidence of these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Children started hemodialysis for end stage renal disease at age of 2 to 16 years will be included in the study.

Exclusion Criteria:

* Patients with known thyroid disease. Patients with a history of autoimmune disease .

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Detection of thyroid function in hemodialysis childern | 6 months
  Detection of decrease thyroid function(T3_T4_TSH) in hemodialysis childern Detection of increase thyroid function(T3_T4_TSH) in hemodialysis childern

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pan B, Du X, Zhang H, Hua X, Wan X, Cao C. Relationships of Chronic Kidney Disease and Thyroid Dysfunction in Non-Dialysis Patients: A Pilot Study. Kidney Blood Press Res. 2019;44(2):170-178. doi: 10.1159/000499201. Epub 2019 Apr 23. PMID 31013508
- [Background] Naseem F, Mannan A, Dhrolia MF, Imtiaz S, Qureshi R, Ahmed A. Prevalence of subclinical hypothyroidism in patients with chronic kidney disease on maintenance hemodialysis. Saudi J Kidney Dis Transpl. 2018 Jul-Aug;29(4):846-851. doi: 10.4103/1319-2442.239646. PMID 30152421